CLINICAL TRIAL: NCT03093714
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate Safety, Pharmacokinetics (PK) and Pharmacodynamics(PD) of FDL169 in Cystic Fibrosis (CF) Subjects Homozygous for the F508del-CFTR Mutation
Brief Title: A Study to Evaluate Safety, PK and PD of FDL169 in Cystic Fibrosis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDL169-2015-04
Record Dates: First submitted 2017-03-16; First posted 2017-03-28 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FDL 169 test formulation (Dose Level 1) (Experimental): Multiple dose (Dose Level 1) FDL 169 test formulation administered as repeat doses in CF subjects
  Interventions: Drug: FDL169
- FDL 169 test formulation (Dose Level 2) (Experimental): Multiple dose (Dose Level 2) FDL 169 test formulation administered as repeat doses in CF subjects
  Interventions: Drug: FDL169
- FDL 169 test formulation ( Dose Level 3) (Experimental): Multiple dose (Dose Level 3) FDL 169 test formulation administered as repeat doses in CF subjects
  Interventions: Drug: FDL169
- Placebo (Placebo Comparator): Multiple dose placebo as repeat doses in CF subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FDL169 — CFTR corrector
  Arms: FDL 169 test formulation ( Dose Level 3); FDL 169 test formulation (Dose Level 1); FDL 169 test formulation (Dose Level 2)
Drug: Placebo — Placebo for FDL169
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, placebo-controlled, dose-escalation study. Enrollment is planned to occur at approximately 14 global sites. Approximately 24 subjects with CF.

DETAILED DESCRIPTION:
This is a multicenter, randomized double-blind, placebo-controlled dose-escalation and parallel-arm, dose-ranging study. Enrollment is planned to occur at approximately 14 global sites. Approximately 24 subjects with CF who are homozygous for the F508del-CFTR mutation will be enrolled in two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a confirmed diagnosis of CF defined as a sweat chloride value ≥60 mmol/L by quantitative pilocarpine iontophoresis or two CF-causing mutations,documented in the subject's medical record or confirmed at screening.
* Age 18 and above on the date of informed consent.
* Weight ≥40 kg.
* Homozygous for the F508del-CFTR mutation. Genotyping to be confirmed at screening.
* Ability to perform a valid, reproducible spirometry test with demonstration of a forced expiratory volume in 1 sec (FEV1) >40% of predicted normal for age, sex and height.
* Screening laboratory tests with no clinically significant abnormalities that would interfere with the study assessments (as judged by the Investigator).
* Subjects who are sexually active must agree to follow the study's contraception requirements.

Exclusion Criteria:

* An acute upper or lower respiratory tract infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 4 weeks prior to Day 1.
* Major complications of lung disease (including massive hemoptysis, pneumothorax, or pleural effusion) within 8 weeks prior to screening.
* Impaired renal function or known portal hypertension.
* History of prolonged QT and/or QTcF (Fridericia's correction) interval (>450 msec) or QTcF >450 msec at Screening.
* History of solid organ or hematological transplantation.
* History of alcohol abuse or drug addiction (including cannabis, cocaine and opiates) during the past year, (as judged by the Investigator).
* Use of ivacaftor or lumacaftor, within 4 weeks of Day 1
* Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for CF or for CF-related conditions within 4 weeks prior to Day 1.
* Ongoing immunosuppressive therapy (including systemic corticosteroids).
* Hemoglobin <10 g/dL.
* Abnormal liver function, at screening.
* Abnormal renal function at screening.
* Ongoing participation in another clinical study or prior participation without appropriate washout (minimum of 10 half- lives or 30 days, whichever is longer) prior to Screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  Safety and tolerability of FDL169 as determined by the incidence of adverse events (AEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Pharmacokinetic parameters, Cmax | 28 days
  The pharmacokinetic parameters of FDL169: maximal plasma concentration (Cmax).
Pharmacokinetic parameters, Tmax | 28 days
  The pharmacokinetic parameters of FDL169: maximal concentration (Tmax).
Pharmacokinetic parameters, AUC | 28 days
  The pharmacokinetic parameters of FDL169: area under the plasma concentration curve (AUC).
Pharmacokinetic parameters, CL/F | 28 days
  The pharmacokinetic parameters of FDL169: clearance (CL/F).
Pharmacokinetic parameters, V/F | 28 days
  The pharmacokinetic parameters of FDL169: apparent volume of distribution (V/F).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Ordonez, MD, Study Chair — Flatley Discovery Lab
Locations (14):
- Australia (3):
  - Mater Misericordiae Ltd, South Brisbane, Queenland
  - The Prince Charles Hospital, Chermside, Queensland
  - The Alfred Hospital, Melbourne
- Czechia (2):
  - FN v Motole, Pediatrická klinika, Centrum cystické fibrózy, Brno
  - FN v Motole, Pediatrická klinika, Centrum cystické fibrózy, Prague
- Germany (4):
  - Charité - Universitätsmedizin Berlin CVK, Berlin
  - Klinik Donaustauf, Zentrum für Pneumologie, Donaustauf
  - Ruhrlandklinik, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
- United Kingdom (5):
  - NICRN Respiratory Research Office, Belfast City Hospital, Belfast
  - Research Dept., Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton Hospital, London
  - The Medicines Evaluation Unit (MEU), Manchester
  - NIHR Wellcome Trust Clinical Research Facility, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662